CLINICAL TRIAL: NCT01990976
Title: Study of Morphology and Functional Magnetic Resonance Imaging (MRI) Muscle Patients With Muscular Dystrophy Type FSHD Benefiting a Physical Training Introduced.
Acronym: FSHD3
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Association Française contre les Myopathies (AFM), Paris (Other); Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: 1208050; 2012-A00430-43 (Other: AFFSAPS)
Record Dates: First submitted 2013-11-18; First posted 2013-11-25 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Muscular Dystrophy; Facioscapulohumeral
Keywords: Muscular Dystrophy; Facioscapulohumeral; Physical training; Magnetic Resonance Imaging; Muscle Biopsy
MeSH Terms: conditions — Muscular Dystrophies | interventions — Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Muscles
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- FSHD training: Only the patients who have participated to the FSHD1 study (NCT01116570) and the FSHD2 study (NCT01689480) can be included in this study.
  Interventions: Device: MRI; Procedure: Biopsy

INTERVENTIONS:
Device: MRI — In Paris centre, a total body NMR imaging will be done with standard T2- and T1-weighted images.
Procedure: Biopsy — biopsy of the vastus lateralis muscle

SUMMARY:
The safety of guided practice of physical activity in myopathies is increasingly accepted, including muscular dystrophies. In facioscapulohumeral dystrophy (FSHD), one of the most common muscular dystrophy, the aerobic training showed its physiological and functional efficiency without affecting the quality of life of patients. The issue of exercise therapy extended to all neuromuscular diseases, as has been rigorously analyzed, shows that the use of a training program combining endurance exercise targeted exercises and strength is even more relevant.

To complete the multidimensional assessments be managed by each team ( physiological assessments, functional tissue and quality of life) it is relevant to continue , for a descriptive study quantitative and qualitative analyzes by muscle imaging and spectroscopy (MRI and Nuclear Resonance Imaging (NMR) spectroscopy ).

DETAILED DESCRIPTION:
These non-invasive assessments already in place at the time of the initial training (FSHD1 study, NCT01116570) will be repeated in the medium (12 months) and long term (30 months) in the same laboratory NMR AIM - CEA , Institute of Myology in Paris (P Carlier ). The data obtained from NMR repeated examinations and those obtained from biochemical analyzes and additional muscle histomorphometric (cellular aging estimation of involution fibroadipose ) on biopsies already programmed (initial, 6 months and 30 months, FSHD2 study, NCT01689480) will be respectively compared to initial time to follow the evolution food and energy capacity of trained muscles. The study of biopsies provide mechanistic arguments and morphometric specific cellular response to exercise, data will be advantageously complemented by NMR specialized examinations extended to all the muscles of the thigh (target of training ) and muscle quantification whole body MRI.

ELIGIBILITY:
Inclusion Criteria:

* Included in the FSHD1 and FSHD2 studies
* Social Security regimen affiliated
* Consent form signed

Exclusion Criteria:

* Severe cardiac or respiratory insufficiency
* Cardiac pacemaker
* Morbid obesity (BMI upper to 35)
* Anti platelet therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with facioscapulohumeral dystrophy and who have participated to the FSHD1 and FSHD2 studies
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2012-05; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Parameters of MRI | 30 months
  whole body imaging T1, T2-weighted

SECONDARY OUTCOMES:
Muscle tissue parameters | 30 months
  muscle biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Léonard FEASSON, MD-PhD, Principal Investigator — CHU de Saint-Etienne
Locations (2):
- France (2):
  - CHU de Grenbole, Grenoble
  - CHU de Saint-Etienne, Saint-Etienne